CLINICAL TRIAL: NCT01863641
Title: The Effect of Calcitriol on Progress and Activity of Lupus Nephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guilan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Amir Maafi, Minister of Student Research Committee, Guilan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1910354604; IRCT2013030912762N1 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2013-05-17; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus nephritis; proteinuria; SLE; calcitriol
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis; Proteinuria | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment group (Experimental): Patients will receive calcitriol at a fixed dose daily.
  Interventions: Drug: calcitriol
- control group (Active Comparator): Patients will receive placebo daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: calcitriol — Patients will receive calcitriol at a fixed dose of 0.25 µg (one oral pearl) daily.
  Arms: treatment group
Drug: placebo — Patients will receive placebo similar to intervention (shape, color and design) 1 oral unit daily.
  Arms: control group

SUMMARY:
The purpose of this study is to determine whether calcitriol is effective in the treatment of lupus nephritis.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease and renal involvement represent one of the most common manifestations of it . On the other hand, there is evidence that vitamin D and its analogs have known immunosuppressant properties and profound effects on glomerular mesangial cell proliferation. Moreover much literature such as animal studies suggests it as a therapeutic intervention in autoimmune disease. The investigators plan to conduct a double blind randomized control clinical trial to study effects of calcitriol on progress and activity of lupus nephritis. Fifty patients with clinically quiescent SLE and biopsy-proven glomerulonephritis will be recruited. They will be treated with calcitriol for 1 year. Proteinuria, renal function, lupus disease activity, serum inflammatory markers will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Baseline Systemic Lupus Erythematosus Disease Activity Index score <= 4
* Estimated glomerular filtration rate more than 15 ml/min/1.73m2
* Proteinuria > 1 g/day (or proteinuria > 1 g/g-Cr) in 2 consecutive samples within 12 weeks despite ACE inhibitor at least 3 months
* On maintenance dose of prednisolone < 15 mg/day with or without other immunosuppressive medications
* Serum calcium level in normal range( 8.5-10.5 mg/dl)
* History of biopsy-proven lupus nephritis clinical quiescent SLE for at least 3 month
* Willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* History of malignancy, including leukemia and lymphoma within the past 2 years; Systemic infection requiring therapy at study entry
* Any other severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* History of drug or alcohol abuse within past 2 years
* Vitamin D deficiency(25 hydroxy vitamin D less than 20ng/ml)
* Participation in any previous trial on vitamin D analogue
* Patients receiving treatment of vitamin D and/or its analogue for other medical reasons within the past 4 weeks
* Patients who are taking multivitamin supplement that contains vitamin D could be enrolled after 4 weeks of wash out period by changing to a preparation that has no vitamin D
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance; Known history of sensitivity or allergy to vitamin D analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
change in proteinuria | baseline and 12 months

SECONDARY OUTCOMES:
risk of lupus flare | baseline and 12 months
change in renal function | baseline and 12 months
  based on the American College of Rheumatology renal response criteria
change in serum inflammatory markers | baseline and 12 months
change in Systemic Lupus Erythematosus Disease Activity Index score | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Banafsheh ghavidel parsa, MD, Study Chair — Guilan University of Medical Sciences, Iran; Alireza Amir Maafi, MD Student, Principal Investigator — Student Research Committee, Guilan University of Medical Sciences, Rasht, Iran
Locations (1):
- Razi hospital, Rasht, Gilan Province, Iran